CLINICAL TRIAL: NCT05672173
Title: Phase 2 Study of the Combination of Lisocabtagene Maraleucel, Nivolumab, and Ibrutinib in Richter's Transformation
Brief Title: Lisocabtagene Maraleucel, Nivolumab and Ibrutinib for the Treatment of Richter's Transformation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22040; NCI-2022-10247 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22040 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Transformed Chronic Lymphocytic Leukemia; Richter Syndrome
MeSH Terms: interventions — Biopsy; Specimen Handling; Cyclophosphamide; fludarabine; ibrutinib; Nivolumab; Blood Component Removal; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, ibrutinib, chemotherapy, liso-cel) (Experimental): Patients receive ibrutinib PO, nivolumab IV, fludarabine IV, cyclophosphamide IV, and liso-cel IV on study. Patients also undergo apheresis, PET/CT, biospecimen collection, and bone marrow biopsy on study. Patients may receive low-moderate intensity chemotherapy in combination with the study induction therapy per treating physician discretion with approval of study principal investigator.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Ibrutinib; Biological: Lisocabtagene Maraleucel; Biological: Nivolumab; Procedure: Pheresis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood specimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and/or aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Biological: Lisocabtagene Maraleucel — Given IV
  Other Names: Anti-CD19-CAR Genetically Engineered Autologous T Lymphocytes JCAR017; Anti-CD19-CAR Genetically Engineered Autologous T-lymphocytes JCAR017; Autologous Anti-CD19-EGFRt-4-1BB-zeta-modified CAR CD8+ and CD4+ T-lymphocytes JCAR017; Breyanzi; JCAR 017; JCAR017
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Procedure: Pheresis — Undergo apheresis
  Other Names: Apheresed; Apheresis; Blood Component Removal; Collection, Apheresis/Leukapheresis; Hemapheresis
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT

SUMMARY:
This phase II trial tests how well adding lisocabtagene maraleucel (liso-cel) to nivolumab and ibrutinib works in treating patients with Richter's transformation. Liso-cel is in a class of medications called autologous cellular immunotherapy, a type of medication prepared by using cells from patient's own blood. It works by causing the body's immune system (a group of cells, tissues, and organs that protects the body from attack by bacteria, viruses, cancer cells and other substances that cause disease) to fight the cancer cells. Nivolumab is in a class of medications called monoclonal antibodies. It works by helping the immune system to slow or stop the grown of cancer. Ibrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals cancer cells to multiply. This helps stop the spread of cancer cells. Giving ibrutinib and nivolumab with Liso-cel may kill more cancer cells in patients with Richter's transformation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the complete response (CR) rate after cycle 3 following lisocabtagene maraleucel (liso-cel) in combination with nivolumab and ibrutinib to treat patients with Richter's transformation (RT).

II. Assess the Unacceptable toxicities (UT) rate within the first 28 days during cycle 1 following liso-cel infusion. (Safety lead-in only)

SECONDARY OBJECTIVES:

I. Assess the safety of liso-cel, nivolumab and ibrutinib to treat patients with RT.

II. Estimate the best CR rate. III. Estimate the best overall response rate (ORR). IV. Estimate duration of response (DOR) at 2 years. V. Assess minimal residual disease (MRD) post liso-cel in participants with CLL at baseline.

VI. Estimate progression free survival (PFS) at 2 years. VII. Estimate overall survival (OS) at 2 years.

EXPLORATORY OBJECTIVES:

I. Evaluate predictive biomarkers of response (genetic and immune) in peripheral blood, apheresis product, infusion product and circulating tumor (ct)DNA.

II. Evaluate the ability of MRD assessed by ctDNA analysis to predict PFS. III. Evaluate changes in the lymph node microenvironment during nivolumab therapy, with an optional pre-CAR T cell infusion lymph node biopsy.

IV. Evaluate the effect of liso-cel on CD19 expression on tumor cells at disease progression.

OUTLINE:

Patients receive ibrutinib orally (PO), nivolumab intravenously (IV), fludarabine IV, cyclophosphamide IV, and liso-cel IV on study. Patients also undergo apheresis, positron emission tomography (PET)/computed tomography (CT), collection of blood samples, and bone marrow biopsy on study. Patients may receive low-moderate intensity chemotherapy in combination with the study induction therapy per treating physician discretion with approval of study principal investigator.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Agreement for confirmatory pre-treatment tumor biopsy

  * If a patient does not have an easily accessible lymph node to biopsy without excessive risk in the opinion of the investigator, archival biopsy material reviewed by a hematopathologist at the enrolling site for study eligibility and baseline correlatives may be acceptable with approval from the Study principal investigator (PI)
* Age: >= 18 years
* Eastern cooperative oncology group (ECOG) <= 2
* Histologically confirmed Richter's Transformation (RT)
* Relapsed / refractory following >=2 prior lines of systemic therapy; OR refractory to first-line chemoimmunotherapy; OR relapsed within 12 months of first line chemoimmunotherapy; OR relapsed after first line of chemoimmunotherapy and not eligible for hematopoietic stem cell transplantation due to comorbidities or age
* Eligible to receive liso-cel and ibrutinib per package inserts
* Fully recovered from the acute toxic effects (except alopecia) to <= Grade 1 to prior anti-cancer therapy
* Absolute neutrophil count (ANC) >= 750/mm^3 unless there is bone marrow involvement
* Platelets >= 75,000/mm^3 unless there is bone marrow involvement
* Total bilirubin =< 1.5 X ULN (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) =< 2.5 x ULN
* Alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* International Normalized Ratio (INR) OR Prothrombin (PT) =< 1.5 x ULN
* Activated Partial Thromboplastin Time (aPTT) =< 1.5 x ULN
* Left ventricular ejection fraction (LVEF) >= 40%

  * Note: To be performed within 28 days prior to Day 1 of protocol therapy.
* Seronegative for HCV*, active HBV (Surface Antigen Negative), and syphilis (RPR)

  * If positive, Hepatitis C RNA quantitation must be performed OR
  * If seropositive for HCV or HBV, nucleic acid quantitation must be performed. Viral load must be undetectable
* Meets other institutional and federal requirements for infectious disease titer requirements

  * Note: Infectious disease testing to be performed within 28 days prior to Day 1 of protocol therapy
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 5 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Subjects who previously received PD1 or PD-L1 inhibitor therapy
* Autologous stem cell transplant within 3 months prior to Day 1 of protocol therapy
* Allogeneic stem cell transplant within 3 months prior to Day 1 of protocol therapy and no active graft versus host disease (GVHD) or need for immunosuppressants
* Chemotherapy, radiation therapy, immunotherapy within 14 days prior to Day 1 of protocol therapy
* Strong CYP3A inducers within 14 days prior to Day 1 of protocol therapy
* Warfarin within 5 days prior to Day 1 of protocol therapy
* Current requirement for oxygen supplementation
* Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. Physiologic replacement of steroids (prednisone =< 7.5 mg /day or equivalent) is allowed throughout the study. Use of "bridging" steroids, to control disease, after leukapheresis and until 3 days prior to CAR T cell infusion, is allowed
* Subjects with lymphoma only involving the central nervous system
* Class III/IV cardiovascular disability according to the New York Heart Association (NYHA) Classification
* Subjects with clinically significant arrhythmia or arrhythmias not stable on medical management within two weeks of screening
* Subjects with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system, including seizure disorder
* Subjects with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 6 months prior to screening
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; non-muscle invasive bladder cancer; malignancy treated with curative intent with no known active disease present for >= 3 years
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Known history of immunodeficiency virus (HIV)
* Females only: Pregnant or breastfeeding
* Subjects with an active, known or suspected autoimmune disease. Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis) not requiring systemic treatment, well controlled asthma and/or mild allergic rhinitis (seasonal allergies) are eligible
* Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | Up to 2 years
  After cycle 3, the rate and associated 95% binomial exact confidence interval will be estimated.
Unacceptable Toxicity (UT) | Up to 28 days post CAR T cell infusion
  Toxicities will be summarized by organ, severity, time of onset and characteristic. UT will be described individually and summarized by count and rate/percentage.

SECONDARY OUTCOMES:
Toxicity | Up to 2 years
  Toxicities will be summarized by organ, severity, time of onset and characteristic. Assessed per ASTCT Consensus Criteria
Best Complete Response (CR) | Up to 2 years
  Defined as the proportion of patients that achieve CR at any time from start of protocol treatment to any disease progression or start of new anticancer treatment.
Overall Response Rate (ORR) | Up to 2 years
  Defined as the proportion of patients that achieve a best response of CR or partial response (PR) from start of protocol treatment prior to any disease progression or start of new anticancer treatment.
Duration of Response (DOR) | Up to 2 years
  Defined as the time from the first documented CR or PR through disease relapse, progression or death. Data for those patients without CR/ PR, disease progression, relapse or death will be captured at last follow up or start of non-protocol anticancer therapy. Those patients that do not achieve CR/PR will be excluded. Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate the DOR.
Minimal Residual Disease (MRD) | Up to 2 years
  Evaluated in the peripheral blood and bone marrow using ClonoSEQ analysis. MRD at baseline will be summarized by descriptive analysis.
Progression Free Survival (PFS) | From start of protocol treatment through disease relapse/ progression or death, assessed up to 2 years
  Data for patients without disease relapse/ progression or death will be collected at the last follow-up or at start of non-protocol anticancer therapy. Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate the PFS.
Overall Survival (OS) | From the start of protocol treatment through death due to any cause, assessed up to 2 years
  Data for alive patients will be collected at last follow up. Kaplan-Meier product limit method with log-log transformation for the confidence interval will be used to estimate the OS.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Siddiqi, Principal Investigator — City of Hope Medical Center
Locations (2):
- United States (2):
  - City of Hope Medical Center, Duarte, California
  - Memorial Sloan Kettering Cancer Center, New York, New York